CLINICAL TRIAL: NCT00872274
Title: An Open Label, Bioequivalence Study of Sumatriptan Succinate 100 mg Tablets (Containing 140 mg of Sumatriptan Succinate Equivalent to 100 mg Sumatriptan) Under Fed Conditions
Brief Title: Bioequivalence Study of Sumatriptan 100mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 220_SUMAT_08
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): sumatriptan succinate tablets 100 mg (containing sumatriptan succinate equivalent to 100 mg of sumatriptan) manufactured by OHM Laboratories In
  Interventions: Drug: sumatriptan 100mg
- 2 (Active Comparator): IMITREX® 100 mg tablets (containing sumatriptan succinate equivalent to 100 mg of sumatriptan)
  Interventions: Drug: sumatriptan 100mg

INTERVENTIONS:
Drug: sumatriptan 100mg

SUMMARY:
To access the single-dose oral bioequivalence of sumatriptan succinate 100 mg tablet (containing 140 mg of sumatriptan succinate equivalent to 100 mg of sumatriptan) of OHM Laboratories Inc. (a subsidiary of Ranbaxy Pharmaceutical Inc. USA) with IMITREX® 100 mg tablet (containing 140 mg of sumatriptan succinate equivalent to 100 mg of sumatriptan) of GlaxoSmithKline in healthy, adult, male, human subjects under fed condition.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomized two-treatment, two-period, two-sequence, single-dose, crossover bioequivalence study comparing sumatriptan succinate tablets 100 mg (containing sumatriptan succinate equivalent to 100 mg of sumatriptan) manufactured by OHM Laboratories Inc. with IMITREX® 100 mg tablets (containing sumatriptan succinate equivalent to 100 mg of sumatriptan) manufactured by GlaxoSmithKline Research Triangle Park NC 27709, Made in Canada in healthy, adult, male, human, subjects under fed conditions.

Following an overnight fast of at least 10 hour, a single oral dose of sumatriptan succinate tablets 100 mg of either test or reference formulation was administered during each period of the study, along with 240 mL of drinking water at ambient temperature under supervision of trained study personnel 30 min after start of a high fat high calorie breakfast.

Thirty-two 32 subjects were enrolled into the study. Twenty-four (24) subjects completed both the periods of the study.

Pharmacokinetic and statistical analyses were performed on data from 24 subjects who completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Were in the age range of 18-45 years.
2. Were neither overweight nor underweight for his height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Had voluntarily given written informed consent to participate in this study.
4. Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.
5. Had a non-vegetarian diet habit.

Exclusion Criteria:

1. Hypersensitivity to Sumatriptan or related group of drugs or to any other drug.
2. History of interment chest pain and or chest tightness which might or might not require medication for relieve.
3. History of headache, vertigo, dizziness with or without nausea vomiting
4. History of intermittent loss of vision
5. History of seizure and or head injury.
6. History of peripheral vascular disease (cramping, tiredness and or severe pain on walking relatively shorter distances persisting on rest, noticeable change in color (blueness or paleness) or temperature (coolness) when compared to the other limb)
7. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
8. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma, head-injury or coma.
9. History of any psychiatric illness, which might impair the ability to provide written informed consent.
10. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
11. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
12. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
13. Presence of values, which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
14. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
15. Clinically abnormal ECG or Chest X-ray.
16. Regular smokers who smoked more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
17. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
18. Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
19. Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
20. Subjects who, through completion of this study, would had donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Ranbaxy Sumatriptan 100mg tablets under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy CPU, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html